CLINICAL TRIAL: NCT00349869
Title: Yoga for Persons With Rheumatoid Arthritis
Brief Title: Yoga for Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: F31AT003362-01A1 (NIH); F31AT003362-01A1 (NIH); R24AT004641 (NIH); Doctoral Dissertation Award (Other: Arthritis Foundation); NCT00346307 (obsolete NCT alias)
Record Dates: First submitted 2006-07-06; First posted 2006-07-10 (Estimated); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Rheumatoid Arthritis; Osteoarthritis
Keywords: inflammatory arthritis; rheumatoid arthritis; knee osteoarthritis; arthritis; yoga
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoarthritis; Arthritis; Osteoarthritis, Knee | interventions — Yoga

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Assessors masked to study condition
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): 8-week yoga program
  Interventions: Behavioral: yoga
- 2 (No Intervention): Usual care control

INTERVENTIONS:
Behavioral: yoga — 8-week yoga program.
  Arms: 1

SUMMARY:
The purpose of this study is to evaluate the impact of yoga on inflammatory arthritis and knee osteoarthritis.

DETAILED DESCRIPTION:
Yoga is a set of ancient Indian theories and practices, focusing on unifying mind, body, and spirit, and promoting strength, balance, and flexibility. The physical aspect of yoga includes poses, breathing techniques, and relaxation. Inflammatory arthritis, a chronic disease characterized by inflammation of the lining of the joints, can cause long-term joint damage, resulting in chronic pain, loss of function, and disability.

The primary objective of this study is to learn how people with inflammatory arthritis and knee osteoarthritis respond to an exercise program of yoga. To accomplish this, 30 persons with inflammatory arthritis or knee osteoarthritis will be randomly assigned to one of two groups. Group one will begin an immediate 8-week program of yoga classes consisting of 60-minute sessions, twice a week. Group two, or the "waitlist" control group, will receive 8 weeks of arthritis education followed by the same 8-week yoga program as group one. Participants also will have blood drawn, and complete various tests. The yoga classes will be taught by an experienced, certified yoga instructor, and are designed especially for the needs of people with inflammatory arthritis and knee osteoarthritis.

This study will provide important data on integrating mind-body activities into the treatment of inflammatory arthritis and knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+ (RA only upper age limit 70)
* Confirmed or probable OA (using pre-specified criteria) OR Rheumatoid arthritis (participation approved by rheumatologist)
* Currently sedentary (physically active for 20 min < 3times/week)

Exclusion Criteria:

* Inability to ambulate without use of assistive device
* Uncontrolled high blood pressure or existing heart condition
* Co-morbid inflammatory condition with overlapping symptoms (i.e., fibromyalgia)
* Surgery within 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2006-08; Primary Completion 2010-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Physical Health | baseline, post intervention, follow-up
  Assessed using SF36 Physical Component Score

SECONDARY OUTCOMES:
Mobility/Fitness | baseline, posttest, follow-up
  Change in flexibility, balance, strength, walk time
RA Disease Activity | baseline, post intervention, follow-up
  DAS28 CRP score
Psychological Function | baseline, , posttest, follow-up
  Change in SF36 MCS, CES-D, PANAS, Perceived Stress and Arthritis Self Efficacy
HRQL | baseline, post intervention, follow-up
  Change in SF36 domains

CONTACTS AND LOCATIONS:
Overall Officials: Susan J. Bartlett, Ph.D., Principal Investigator — Associate Professor of Medicine, Johns Hopkins Rheumatology
Locations (1):
- Johns Hopkins Arthritis Center, 5501 Hopkins-Bayview Circle, Ste 1B.14, Baltimore, Maryland, United States

REFERENCES:
- [Result] Bartlett SJ, Moonaz SH, Mill C, Bernatsky S, Bingham CO 3rd. Yoga in rheumatic diseases. Curr Rheumatol Rep. 2013 Dec;15(12):387. doi: 10.1007/s11926-013-0387-2. PMID 24173693
- [Result] Haaz S, Bartlett SJ. Yoga for arthritis: a scoping review. Rheum Dis Clin North Am. 2011 Feb;37(1):33-46. doi: 10.1016/j.rdc.2010.11.001. Epub 2010 Dec 3. PMID 21220084
- [Result] Haaz S, Bingham CO, Bathon JM, Bartlett SJ. The effect of yoga on clinical parameters in patients with rheumatoid arthritis. Arthritis & Rheumatism 2008;58:S893-S4.
- [Result] Haaz S, Bingham III CO, Bartlett SJ. Adherence to an 8-week yoga program for RA and OA: Who drops out and why? Arthritis & Rheumatism 2009;60:1978.
- [Result] Moonaz SH, Bingham CO 3rd, Wissow L, Bartlett SJ. Yoga in Sedentary Adults with Arthritis: Effects of a Randomized Controlled Pragmatic Trial. J Rheumatol. 2015 Jul;42(7):1194-202. doi: 10.3899/jrheum.141129. Epub 2015 Apr 1. PMID 25834206
- See also: Yoga for Arthritis — http://www.hopkinsarthritis.org/patient-corner/disease-management/yoga-for-arthritis/